CLINICAL TRIAL: NCT06760533
Title: Pilot Proof of Concept Study Evaluating the Potential Psilocybin Assisted Psychotherapy (PAP) as a Therapeutic Tool for Patients Suffering From Severe Irritable Bowel Syndrome.
Brief Title: Psilocybin-Assisted Psychotherapy in Treating Irritable Bowel Syndrome (IBS)
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-00001
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Psilocybin; Niacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention: Psilocybin (Experimental): Participants assigned to the intervention arm will receive psilocybin.
  Interventions: Drug: Psilocybin 25 mg; Behavioral: Psychotherapy Treatment Session
- Control: Niacin (Placebo) (Placebo Comparator): Participants assigned to the control arm will receive a placebo (niacin).
  Interventions: Behavioral: Psychotherapy Treatment Session; Drug: Niacin 100 mg

INTERVENTIONS:
Drug: Psilocybin 25 mg — Psilocybin 25 mg (active treatment) administered during the psychotherapy treatment session.
  Arms: Intervention: Psilocybin
Behavioral: Psychotherapy Treatment Session — The psychotherapy treatment sessions will be conducted by two therapists, who will be both present for all the sessions during three phases of treatment: Preparation, Medication Administration, and Integration.
Drug: Niacin 100 mg — Niacin 100 mg (placebo) administered during the psychotherapy treatment session.
  Arms: Control: Niacin (Placebo)

SUMMARY:
This study will serve as a pilot randomized controlled trial to assess the feasibility of Psilocybin-Assisted Psychotherapy (PAP) in Treating Irritable Bowel Syndrome (IBS). Patients with severe IBS will undergo 3 pre-psychotherapy sessions with two licensed and trained psychedelic therapists, then will be randomized to undergo a guided psychotherapy session with single 25 mg oral "high" dose of psilocybin or a single 100 mg dose of niacin (active placebo) and attend 4 post-therapy integration sessions.

ELIGIBILITY:
Inclusion Criteria:

* Severe IBS patients meeting Rome IV criteria. Severe IBS is defined by IBS-SS >300, or one or more emergency room (ER) visit for abdominal pain in the last year.
* Experiencing persistent IBS symptoms despite pharmacologic therapy
* Have an identified support person
* Agree to be accompanied home (or to an otherwise safe destination) by the support person, or another responsible party, following dosing
* Participants of childbearing potential must agree to practice an effective means of birth control throughout the duration of the study.
* Participants must agree to send outside medical records in order for the study team to verify eligibility.

Exclusion Criteria:

* Unstable medical conditions or serious abnormalities on complete blood count, chemistries, or ECG that in the opinion of the study physician would preclude safe participation in the trial. Some examples include:

  * Congestive heart failure
  * Clinically significant arrhythmias (e.g.,
  * Ventricular fibrillation, torsades) or clinically significant ECG abnormality (i.e., corrected QT interval > 450)
  * Recent acute myocardial infarction or
  * Evidence of ischemia (in the last year)
  * Malignant hypertension
  * Congenital long QT syndrome
  * History of valvular heart disease
  * Acute renal failure
  * Moderate to Severe hepatic impairment (Child Pugh class B and C).
  * Respiratory failure
  * Recent stroke (< 1 year from signing of consent)
  * Laboratory tests abnormalities (ALT ≥ 2X upper limit of normal (ULN), aspartate aminotransferase (AST) ≥ 2X ULN, Hemoglobin<11.5, platelets <150, White Blood Cells (WBC)>10, Sodium>150, Potassium K<3.5 or K>5.2)
  * Abnormal and clinically significant results on the physical examination (BP>139/89 mmHG), heart rate (HR)>90bpm,
  * History of Pulmonary hypertension
* Significant central nervous system (CNS) pathology. Examples include:

  * Primary or secondary cerebral neoplasm
  * Epilepsy
  * History of stroke
  * Cerebral aneurysm
  * Dementia
  * Delirium
* Primary psychotic or affective psychotic disorders. Examples include current or past DSM-5 criteria for:

  * Schizophrenia spectrum disorders
  * Schizoaffective disorder
  * Bipolar I or II disorder with psychotic features
  * Major Depressive Disorder
  * Substance induced psychotic disorders
  * Paranoid personality disorder
  * Delusional disorder
  * Borderline personality disorder
  * Any other psychotic illness
* Family history of psychotic or serious bipolar spectrum illnesses. Examples include first-degree relative with:

  * Schizophrenia spectrum disorders
  * Schizoaffective disorder
  * Bipolar I disorder with psychotic features
  * Any other psychotic illness
* High risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation. Examples include:

  * Agitation
  * Violent behavior
* Active substance use disorders (SUDs) defined as Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for moderate or severe alcohol or drug use disorder (excluding caffeine and nicotine) within the past year
* Clinically significant suicidality or high risk of completed suicide defined as:

  * 'Yes' to C-SSRS Suicidal Ideation items 4 or 5 within the last 2 months at Screening or 'since last visit' at Baseline
  * Any C-SSRS Suicidal Behavior item within the past 12 months at Screening or 'since last visit' at Baseline, as defined by 'Yes' to any of the following on the C-SSRS: actual attempt, interrupted attempt, aborted attempt, or preparatory acts
  * Have any suicidal ideation or thoughts, in the opinion of the study physician or PI, that presents a serious risk of suicidal or self-injurious behavior
* History of hallucinogen persisting perception disorder (HPPD)
* Pregnancy/lactation
* Cognitive impairment as defined by: Montreal Cognitive Assessment Test (MoCA) < 23
* Concurrent Medications

  * Antidepressants
  * Centrally-acting serotonergic agents (e.g., monoamine oxidase inhibitors (MAOIs))
  * Antipsychotics (e.g., first and second generation)
  * Mood stabilizers (e.g., lithium, valproic acid)
  * Aldehyde dehydrogenase inhibitors (e.g., disulfiram)
  * Significant inhibitors of UGT 1A0 or UGT 1A10
  * Niacin
* Subjects should not also be taking serotonin-acting dietary supplements (such as 5-hydroxy-tryptophan or St. John's wort)
* Have a positive urine drug test including Amphetamines, Barbiturates, Buprenorphine, Benzodiazepines, Cocaine, Methamphetamine, 3,4-methylenedioxymethamphetamine (MDMA), Methadone, Opiates (Morphine, Oxycodone), Phencyclidine (PCP)
* Have a psychiatric condition judged to be incompatible with establishment of rapport with the study therapists or safe exposure to psilocybin
* Have any psychological or physical symptom, medication or other relevant finding prior to randomization, based on the clinical judgment of the PI or relevant clinical study staff that would make a participant unsuitable for the study.
* Have an allergy or intolerance to either psilocybin on Niacin
* Be enrolled in another clinical trial assessing intervention(s) for anxiety, depression, and/or existential distress (e.g., pharmacologic or psychotherapeutic interventions)
* Are unable to provide external medical records or refuse to provide external medical records.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Abdominal Pain Severity Numeric Rating Scale (APS-NRS) Score | Baseline, Week 6
  A single-item assessment of abdominal pain severity in patients with IBS. Patients rate their pain severity on a scale from 0 (no pain) to 10 (worst possible pain). The total score ranges from 0-10; lower scores indicate less severe pain.

SECONDARY OUTCOMES:
Change in IBS Severity Scoring System (IBS-SSS) Score | Baseline, Week 6
  The IBS-SSS asks five questions about the severity of IBS symptoms over the past 10 days: abdominal pain, abdominal distention, bowel habits, and quality of life. Each question is rated on a 100-point scale. The total score is the sum of responses and ranges from 0-500; lower scores indicate less severe symptoms, where 75-175 = mild; 175-300 = moderate; and greater than 300 = severe.
Hospital Anxiety and Depression Scale: Anxiety Score | Baseline, Week 6
  The Hospital Anxiety and Depression Scale asks 14 questions related to anxiety and depression. The Anxiety subscale comprises 7 questions; each are rated on a scale from 0-3. The total Anxiety score ranges from 0-21; higher scores indicate more severe anxiety.
Hospital Anxiety and Depression Scale: Depression Score | Baseline, Week 6
  The Hospital Anxiety and Depression Scale asks 14 questions related to anxiety and depression. The Depression subscale comprises 7 questions; each are rated on a scale from 0-3. The total Depression score ranges from 0-21; higher scores indicate more severe depression.
Number of Participants with "Type 3" or "Type 4" Rating on Bristol Stool Form Scale | Baseline
  The Bristol Stool Form Scale rates the consistency of stool on the following scale:
  Type 1 and 2: May be difficult to pass, may indicate constipation. Type 3 and 4: Ideal stools. Type 5: Trending toward diarrhea. Type 6 and 7: Diarrhea.
  This measure assesses the number of participants with Type 3 and 4 (ideal) stools.
Number of Participants with "Type 3" or "Type 4" Rating on Bristol Stool Form Scale | Month 6
  The Bristol Stool Form Scale rates the consistency of stool on the following scale:
  Type 1 and 2: May be difficult to pass, may indicate constipation. Type 3 and 4: Ideal stools. Type 5: Trending toward diarrhea. Type 6 and 7: Diarrhea.
  This measure assesses the number of participants with Type 3 and 4 (ideal) stools.

CONTACTS AND LOCATIONS:
Overall Officials: Maysaa El Zoghbi, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be made available to other researchers.